CLINICAL TRIAL: NCT02612727
Title: Filtered Sunlight Phototherapy to Treat Significant Jaundice: Safety and Efficacy in Neonates
Acronym: FSPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1108M03601_Phase 2
Record Dates: First submitted 2015-10-20; First posted 2015-11-24 (Estimated); Results first posted 2019-06-19 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-06

CONDITIONS: Jaundice, Neonatal
Keywords: Hyperbilirubinemia, Neonatal
MeSH Terms: conditions — Jaundice, Neonatal; Hyperbilirubinemia, Neonatal

STUDY DESIGN:
Intervention Model Description: Non-inferiority trial comparing the two methods of phototherapy
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Filtered-sunlight phototherapy (Experimental): Infants will receive >= four hours per day of filtered-sunlight phototherapy for 1 to 10 days. The filtering will be done using Air Blue 80 window tinting film.
  Interventions: Device: Filtered-sunlight phototherapy
- Intensive phototherapy (Active Comparator): Infants will receive >= four hours per day of intensive phototherapy for 1 to 10 days.
  Interventions: Device: Intensive phototherapy

INTERVENTIONS:
Device: Filtered-sunlight phototherapy — Infants will receive >= four hours per day of filtered-sunlight phototherapy for 1 to 10 days. The filtering will be done using Air Blue 80 window tinting film.
  Arms: Filtered-sunlight phototherapy
Device: Intensive phototherapy — Infants will receive >= four hours per day of intensive phototherapy for 1 to 10 days.
  Arms: Intensive phototherapy

SUMMARY:
At present, much of sub-Saharan Africa, including Nigeria and other resource-limited countries, are without ready access to CPT, due to factors including the lack of PT devices, which are expensive and require consistent electric power to operate. NHB is a significant cause of neonatal morbidity and mortality, but preventable when appropriate treatment is initiated. We have shown that FS-PT is safe and efficacious for the treatment of mild-moderate NHB. The major goal of this study is to demonstrate that FS-PT is efficacious for the treatment of significant/severe NHB, generally defined as TB of ≥12-14mg/dL (but more specially as defined as needing phototherapy per American Academy of Pediatric 2004 guidelines). This arm was done at 1 site in Nigeria (in Ogbomoso). The rationale for conducting the study is that in Nigeria, and other countries that cannot afford effective commercial light devices and/or have no reliable electric power to operate them, filtered sunlight phototherapy might offer a safe and effective treatment for neonatal jaundice.

DETAILED DESCRIPTION:
Severe neonatal hyperbilirubinemia (NHB) and its progression to kernicterus is a leading cause of deaths and disabilities among newborns in the developing world, particularly in sub-Saharan Africa including Nigeria. Many infants live in villages/towns far from clinical facilities capable of providing conventional artificial blue light phototherapy (CPT) which is the standard treatment for NHB in the industrialized world. Hence, more babies succumb to this preventable tragedy principally on account of lack of electricity and/or available/affordable CPT.

To make treatment of NHB more readily available, we designed and tested a novel, yet simple, practical alternative device to deliver blue light PT in underserved areas from filtered sunlight. The investigators pilot study demonstrated that appropriately filtered sunlight phototherapy (FS-PT) not only offers safe and affordable treatment for infants with mild-moderate NHB, but is also no less efficacious than CPT. Other studies have shown faster decline at higher bilirubin (TB) levels and with higher irradiances. The next logical step to move this urgently needed and exciting therapy forward is to test FS-PT in infants with significant/severe NHB as defined by the American Academy of Pediatrics (AAP) criteria for high-risk infants. In doing so, the investigators will potentially be preventing acute bilirubin encephalopathy (ABE) and kernicterus in many of these infants.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be eligible to participate in the study if all of the following conditions exist:

  1. At time of birth, infant is > 35 weeks gestation (or ≥ 2.2 kg if gestational age is not available.
  2. Infant is < 14 days old at the time of enrollment.
  3. Infant has an elevated TB defined as at the level recommended for high-risk infants per AAP guidelines or higher.
  4. Parent or guardian has given consent for the infant to participate.

Exclusion Criteria:

* Subjects will be excluded from enrollment in the study if any of the following conditions exist:

  1. Infants with a condition requiring referral for treatment not available at the hospital study site.
  2. Infants with a life-expectancy of < 24 hours at screening enrollment.
  3. Infants requiring oxygen therapy unless that can be provided while under PT.
  4. Infants clinically dehydrated or sunburned at the time of screening enrollment.
  5. Infants with a temperature < 36.0 or > 37.5 degrees Centigrade that does not return to normothermia within 1 hour.

Max Age: 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 174 (Actual)
Dates: Start 2012-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tina M Slusher, Principal Investigator — University of Minnesota
Locations (1):
- Bowen University Teaching Hospital, Ogbomoso, Nigeria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olusanya BO, Omololu OM, Osamebor FB, Olufosoye A, Alo T, Olaifa SM, Emokpae AA, Olusanya JO, Mabogunje CA. Filtered-sunlight phototherapy for newborns with moderate-to-severe hyperbilirubinemia: a randomized trial. Pediatr Res. 2025 Jun 28. doi: 10.1038/s41390-025-04207-6. Online ahead of print. PMID 40581699
- [Derived] Olusanya BO, Emokpae AA, Aina OA, Imam ZO, Olaifa SM, Owolabi OB, Osamebor FB, Olufosoye A, Alo T, Osadolor A Jr, Olusanya JO, Mabogunje CA. Heliotherapy for neonates with severe-to-hazardous hyperbilirubinemia: a randomized controlled, non-inferiority trial. Sci Rep. 2024 Oct 27;14(1):25646. doi: 10.1038/s41598-024-77085-3. PMID 39465350

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Filtered-sunlight Phototherapy | Intensive Phototherapy
Started | 87 | 87
Completed | 82 | 83
Not Completed | 5 | 4
Not completed — Parent request | 4 | 1
Not completed — Needed treatment incompatible with PT | 1 | 1
Not completed — Direct hyperbilirubinemia | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Filtered-sunlight Phototherapy | Intensive Phototherapy | Total
Number analyzed (Participants) | 87 | 87 | 174
Age, Continuous [Median (Inter-Quartile Range); unit: hours] | 47 [27 to 102] | 59 [33 to 114] | 57 [29 to 112]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex information was missing for one infant in each group.
  Participants
    number analyzed (Participants) | 86 | 86 | 172
    Female | 34 | 30 | 64
    Male | 52 | 56 | 108

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Phototherapy
Description: For a given evaluable treatment day, the phototherapy treatment was deemed effective if that infant on that day had a decrease in serum bilirubin level or (if <72hrs old) an rate of increase of less than 0.2 mg/dL/h. Therefore efficacy is reported as a percentage of the evaluable treatment days (i.e. number of effective evaluable treatment days divided by total number of evaluable treatment days).
Time Frame: 2 to 10 days
Population: The efficacy analysis used all treatment days where an infant received >=4h of PT and both bilirubin levels were available. 87 infants received 215 treatment days of FSPT, but only 133 of those days (in 79 infants) were analyzable for efficacy. Similarly, 87 infants received 219 days of IntPT, but only 152 days (in 83 infants) were analyzable.
Measure: Count of Units; unit: treatment days
Units Other Than Participants: treatment days
Arm/Group | Filtered-sunlight Phototherapy | Intensive Phototherapy
Number analyzed (Participants) | 79 | 83
Number analyzed (treatment days) | 133 | 152
treatment days | 116 | 135

2. Primary Outcome: Safety of Phototherapy
Description: For a given treatment day, the phototherapy treatment was deemed safe if that infant on that day did not have to be withdrawn from treatment due to hypo- or hyperthermia, sunburn or dehydration. Therefore safety is reported as a percentage of the total treatment days (i.e. number of safe treatment days divided by total number of treatment days).
Time Frame: 2 to 10 days
Measure: Count of Units; unit: treatment days
Units Other Than Participants: treatment days
Arm/Group | Filtered-sunlight Phototherapy | Intensive Phototherapy
Number analyzed (Participants) | 87 | 87
Number analyzed (treatment days) | 215 | 219
treatment days | 215 | 219

ADVERSE EVENTS:
Arm/Group | Filtered-sunlight Phototherapy | Intensive Phototherapy
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/87
Other Adverse Events (participants affected / at risk) | 0/87 | 0/87

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No